CLINICAL TRIAL: NCT01781728
Title: Phase II Study to Evaluate Stereotactic Body Radiation Therapy For Palliative Management of Unresectable Recurrent or Residual Pancreatic or Periampullary Adenocarcinoma
Brief Title: Palliative Stereotactic Radiation for Pancreatic or Periampullary Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1273; NA_00070233 (Other: JHMIRB)
Record Dates: First submitted 2012-08-08; First posted 2013-02-01 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer; Periampullary Adenocarcinoma
Keywords: recurrent; unresectable; residual; stereotactic body radiation therapy (SBRT); palliative management
MeSH Terms: conditions — Pancreatic Neoplasms; Recurrence | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, controlled Phase 2 trial
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Locally advanced pancreatic cancer or locally recurrent pancreatic ductal adenocarcinoma (Experimental): Patients with pathologically confirmed, locally advanced pancreatic ductal adenocarcinoma (LAPC), unresectable at diagnosis, or local recurrence pancreatic ductal adenocarcinoma (PDAC) after prior surgical resection.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Stereotactic Body Radiation Therapy (SBRT) which included 5 consecutive fractions of 25 to 33 Gy, following 3 months of multiagent chemotherapy.

SUMMARY:
The investigators are looking to see if a certain dose of stereotactic body radiation therapy (SBRT) may be a viable treatment option for recurrent or residual pancreatic or periampullary adenocarcinoma.

DETAILED DESCRIPTION:
No standard treatment option has yet been established for patients with recurrent or residual disease after definitive treatment of pancreatic or periampullary cancers (duodenal, ampullary, bile duct). Linac based stereotactic body radiation therapy (SBRT) administered in 1-3 fractions has been shown to be an effective treatment option for patients with unresectable, locally advanced pancreatic adenocarcinoma, achieving local control rates of 84-92% at one year. Associated late gastrointestinal toxicity rates have been reported to be 22-25% at 1 year. We hypothesize that similarly excellent local control rates (80-90% at one year) with a reasonable rate of toxicity (≤20%) can be achieved using Linac based SBRT delivered as 5 Gy x 5 for patients with local failure (remaining disease) after previous treatment with conventional chemoradiation therapy (CRT) with or without surgery and as 6.6 Gy x 5 for radiation-naïve patients with local failure (remaining disease) after previous treatment with surgery and/or chemotherapy. The toxicities of note for this trial are grade 2 and greater gastritis, fistula, enteritis, ulcer, or any other grade 3 or greater gastrointestinal toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Karnofsky Performance Status greater than or equal to 70%
* confirmed pancreatic or periampullary adenocarcinoma
* pancreatic or periampullary tumor less than 8.0 cm in greatest axial dimension
* Either:

  * standard of care treatment for pancreatic cancer that included radiation therapy

    * patients may be receiving continued chemotherapy post initial CRT. or
  * standard of care treatment for pancreatic cancer that did not include radiation therapy * patients must have attempted chemotherapy upon initial diagnosis
* acceptable organ and marrow function as determined by blood tests
* ability to understand and give consent
* must be a patient to be treated with SBRT only at Johns Hopkins Hospital
* life expectancy of greater than 3 months

Exclusion Criteria:

* extensive metastatic disease
* performance status of less than 70
* children are excluded form the study
* no uncontrolled intercurrent illness
* no concurrent malignancy other than melanoma
* pregnant or breast feeding women are excluded
* women who are not post-menopausal and have a positive pregnancy test
* life expectancy of less than 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Started | 48
Completed (45 patients were followed until death and 3 patients were still alive at last follow-up) | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Late Gastrointestinal Toxicities
Description: Late (Up to 3 months post-treatment to date of first progression or date of death, (whichever comes first-up to 36 months) Grade 2 or greater gastritis, enteritis, fistula, or ulcer and any other grade 3 or greater gastrointestinal toxicity attributable to Stereotactic Body Radiation Therapy (SBRT).
  Toxicity was assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 4.0) and the Radiation Therapy Oncology Group radiation morbidity scoring criteria.
Time Frame: 3 months post-treatment to date of first progression or date of death, whichever comes first assessed up to 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma: Stereotactic Body Radiation Therapy (SBRT): 6.6 Gy x 5 (over 1-2 weeks)*
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 48
Participants | 13

2. Secondary Outcome: Acute Gastrointestinal Toxicity
Description: Any acute gastrointestinal (GI) toxicities grade 3 or greater.
Time Frame: within 3 months of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma: Patients with pathologically confirmed, locally advanced pancreatic ductal adenocarcinoma (LAPC), unresectable at diagnosis, or local recurrence pancreatic ductal adenocarcinoma (PDAC) after prior surgical resection.
  Stereotactic Body Radiation Therapy (SBRT): Stereotactic Body Radiation Therapy (SBRT) which included 5 consecutive fractions of 25 to 33 Gy.
  Chemotherapy drug: 3 months of multiagent chemotherapy
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 48
Participants | 3

3. Secondary Outcome: Local Progression Free Survival From SBRT
Description: Local progression free survival defined as the length of time (months) during and after the treatment of a disease that a patient lives with cancer, but the disease does not worsen.
Time Frame: From date of randomization until the date of first documented progression or death from any cause (up to 36 months).
Measure: Median (95% Confidence Interval); unit: Months until local progression
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 48
Months until local progression | 14.6 [11.6 to 23]

4. Secondary Outcome: Local Progression Free Survival From Diagnosis
Description: as for outcome 3
Time Frame: From date documented diagnosis to date of first documented local disease progression.
Measure: Median (95% Confidence Interval); unit: Months until local progression
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 48
Months until local progression | 21.6 [16 to 29.7]

5. Secondary Outcome: Change in Patient Reported Quality of Life (PR-QOL) Assessment at Baseline (Pre-treatment) and 3 Months (Post-Treatment)
Description: To evaluate whether a change in patient reported quality of life (QoL) occurred between baseline (pre-SBRT) and at 3 months (post-SBRT) using the European Organization for Research and Treatment in Cancer quality of life core cancer questionnaire with the pancreatic cancer module (EORTC QLQ-C30/Pan26). This assessment is a multi-dimensional, 30-item questionnaire which assesses 5 functional scales (physical, role, cognitive, emotional and social), 3 symptom scales ( fatigue, pain and nausea/vomiting), a global health/QoL scale as well as 6 single items. There are also 26 questions specific to patients with pancreatic cancer.
  Scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Time Frame: Baseline (Pre-SBRT) and at 3 months (Post-SBRT)
Population: Not all patients completed the QOL assessments. In this case 43 of the 48 patients completed assessments.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 43
score on a scale | 0 [-10 to 10]

6. Secondary Outcome: Linear Accelerator (Linac) Based SBRT Pain Control
Description: To evaluate the ability of Linac based SBRT to provide pain control among symptomatic patients as measured by pain medication requirement at 3, 6 and 12 months after treatment.
Time Frame: 3, 6, and 12 months after treatment
Population: We prioritized collecting and analyzing data for the primary outcome of this study which is reported in ClinicalTrials.gov. Unfortunately, due to lack of funding, we were not able to collect and analyze all secondary outcome data as planned.
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 0

7. Secondary Outcome: Linac Based SBRT Standardization
Description: To develop and standardize Linac based SBRT delivery and dosimetric parameters
Time Frame: 3, 6, and 12 months after treatment
Population: We prioritized collecting and analyzing data for the primary outcome of this study which is reported in ClinicalTrials.gov. Unfortunately, due to lack of funding, we were not able to collect and analyze all secondary outcome data as planned. Therefore, dosimetric parameters were not developed
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 0

8. Secondary Outcome: FDG-PET Use for Planning and Estimation of Survival
Description: To evaluate the utility of FDG-PET for treatment planning and estimation of progression-free survival.
Time Frame: 3, 6, and 12 months after treatment and then annually thereafter
Population: as for outcome 6
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 0

9. Secondary Outcome: Toxicity for Patients With Chemotherapy, Surgery (Resection) and Radiation for Tumor Assessments
Description: Toxicity was assessed for grade ≥2 gastrointestinal toxic effects using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0) and the Radiation Therapy Oncology Group radiation morbidity scoring criteria.
Time Frame: Up to 36 months
Population: Participants who had chemotherapy, surgery (resection) and radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 13
Participants | 6

10. Secondary Outcome: Toxicity for Patients With Chemotherapy and Radiation (no Resection)
Description: as for outcome 9
Time Frame: Up to 36 months
Population: Participants who had chemotherapy and radiation (no resection)
Measure: Count of Participants; unit: Participants
Groups:
- Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma: Patients with locally advanced pancreatic ductal adenocarcinoma (LAPC), unresectable at diagnosis, or local recurrence pancreatic ductal adenocarcinoma (PDAC) after prior surgical resection.
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
Number analyzed (Participants) | 13
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma
All-Cause Mortality (participants affected / at risk) | 45/48
Serious Adverse Events (participants affected / at risk) | 10/48
Other Adverse Events (participants affected / at risk) | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma (N=48)
Duadenal Ulcer (Gastrointestinal disorders) | 1 (1)
Liver Abcess (Hepatobiliary disorders) | 1 (3)
Enteritis (Hepatobiliary disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (2) — Grade 4
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) — Grade 3
Vomiting/Pain (General disorders) | 1 (1)
Biliary Obstruction (Gastrointestinal disorders) | 1 (1)
Fistula (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Locally Advanced Pancreatic Cancer or Locally Recurrent Pancreatic Ductal Adenocarcinoma (N=48)
Ulcer (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT01781728/Prot_SAP_000.pdf